CLINICAL TRIAL: NCT05467332
Title: Invasive Measurement of Positive Tracheal Pressure Generated by High Flow Nasal Oxygen Administration in Critically Ill Patients After Extubation: a Physiologic Study.
Brief Title: Tracheal Positive Pressure During High Flow Nasal Oxygen Administration in Critically Ill Patients: a Physiologic Study.
Acronym: HPEEP
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Azienda Sanitaria-Universitaria Integrata di Udine (Other)
Responsible Party: Principal Investigator, Cristian Deana, Medical Doctor, Anesthesiologist and Critical Care Physician, Azienda Sanitaria-Universitaria Integrata di Udine
Other Study IDs: HPEEP
Record Dates: First submitted 2022-07-18; First posted 2022-07-20 (Actual); Last update posted 2023-01-31 (Actual); Status verified 2023-01

CONDITIONS: Acute Respiratory Failure; High Flow Nasal Cannula; Critically Ill; Airway Disease; Positive End Expiratory Pressure; Diaphragm Disease
Keywords: intensive care unit, critically ill patient, high flow nasal cannula, PEEP, respiratory failure, non invasive ventilation
MeSH Terms: conditions — Critical Illness; Respiratory Insufficiency

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- CRITICALLY ILL PATIENTS: CRITICALLY ILL PATIENTS AFTER INVASIVE MECHANICAL VENTILATION READY TO BE EXTUBATED.
  Interventions: Device: HIGH FLOW NASAL OXYGEN

INTERVENTIONS:
Device: HIGH FLOW NASAL OXYGEN — BEFORE EXTUBATION, AN AIRWAY EXCHANGE CATHETER (AEC) WILL BE PUT INTO THE PATIENTS' TRACHEA AND IT WILL REMAIN IN SITE AFTER EXTUBATION. THROUGH AN AEC CONNECTED TO A PRESSURE MONITOR, IT WILL BE RECORDED TRACHEAL PRESSURE DURING SPONTANEOUSLY BREATHING PATIENT AT DIFFERENT FLOW RATES OF HFNC THAT WILL BE APPLIED JUST AFTER EXTUBATION.
  MEANWHILE, VITAL PARAMETERS RECORDED WITH A MULTIPARAMETRIC MONITOR WILL BE RECORDED.
  FINALLY, MONITORING OF ELECTRICAL ACTIVITY OF DIAPHRAGM WILL BE RECORDED THROUGH A DEDICATED NASOGASTRIC TUBE TO EVALUATE IT AT DIFFERENT FLOW RATES.
  Other Names: AIRVO2, FISHER&PAYKEL

SUMMARY:
High flow nasal cannula administration in critically ill patients is frequently used to improve acute respiratory failure or to prevent respiratory failure after extubation.

It acts generating a mild positive pressure in the airways and by reducing respiratory effort of patients.

However to the best of our knowledge, no study to date has directly measured the amount of positive pressure generated in the trachea of patients.

The primary aim, therefore, of this study measures this positive pressure after extubation in critically ill patients.

ELIGIBILITY:
Inclusion Criteria: CRITICALLY ILL PATIENTS AFTER MECHANICAL VENTILATION LASTED AT LEAST 72 HOURS

* age 18-80 years

Exclusion Criteria:

* COPD stage >1 according to GOLD classification
* end stage organ disease (liver, kidney, heart, lung)
* neuromuscular disease
* neoplasm
* previous tracheostomy
* obesity with BMI > 35 Kg/m2
* non collaborative patient

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: CRITICALLY ILL PATIENTS REQUIRING INVASIVE MECHANICAL VENTILATION FOR AT LEAST 72 HOURS AND READY FOR EXTUBATION.
Sampling Method: Non-Probability Sample
Enrollment: 20 (Estimated)
Dates: Start 2023-04 (Estimated); Primary Completion 2023-09 (Estimated); Study Completion 2023-12 (Estimated)

PRIMARY OUTCOMES:
HFNC-PEEP | 3 HOURS
  THE LEVEL OF POSITIVE AIRWAY PRESSURE GENERATED BY DIFFERENT FLOW RATES OX OXYGEN WILL BE RECORDED.
  FLOW RATE STARTS AT 10 L/MIN AND IT WILL BE INCREASED A 10 L/MIN STEP EVERY 30 MINUTES UNTIL 60 L/MIN.

SECONDARY OUTCOMES:
HFNC-EADI | 3 HOURS
  ELECTRICAL ACTIVITY OF THE DIAPHRAGM WILL BE RECORDED THROUGH A DEDICATED NASOGASTRIC TUBE DURING ALL THE PROCESS.
  FLOW RATE STARTS AT 10 L/MIN AND IT WILL BE INCREASED A 10 L/MIN STEP EVERY 30 MINUTES UNTIL 60 L/MIN.

CONTACTS AND LOCATIONS:
Overall Officials: Cristian Deana, MD, Principal Investigator — Health Integrated Agency of Friuli Centrale, via Pozzuolo 330, 33100 Udine, Italy
Locations (1):
- Cristian Deana, Udine, Italy

IPD SHARING:
Plan to Share IPD: No